CLINICAL TRIAL: NCT00889486
Title: A Multicenter, Randomized, Double-Blind, Placebo-Controlled, Parallel-Group, Phase 2 Evaluation of the Safety and Efficacy of Once-Daily Administrations of TZP 102 for the Treatment of Symptomatic Gastroparesis in Patients With Diabetes Mellitus
Brief Title: Safety and Efficacy of Once-daily Oral Administrations of TZP-102 for Gastroparesis in Patients With Diabetes Mellitus
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Tranzyme, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: TZP-102-CL-G002
Record Dates: First submitted 2009-04-28; First posted 2009-04-29 (Estimated); Last update posted 2012-12-11 (Estimated); Status verified 2012-12

CONDITIONS: Gastroparesis; Diabetes Mellitus
Keywords: gastroparesis; diabetes mellitus; delayed gastric emptying
MeSH Terms: conditions — Gastroparesis; Diabetes Mellitus

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: No

ARMS (4):
- Placebo (Placebo Comparator): Four placebo capsules taken orally once per day for 28 days
  Interventions: Drug: Placebo
- 10 mg TZP-102 (Experimental): One 10 mg TZP-102 Capsule and three placebo capsules taken orally once per day for 28 days
  Interventions: Drug: TZP-102; Drug: Placebo
- 20 mg TZP-102 (Experimental): Two 10 mg TZP-102 Capsules and two placebo capsules taken orally once per day for 28 days
  Interventions: Drug: TZP-102; Drug: Placebo
- 40 mg TZP-102 (Experimental): Four 10 mg TZP-102 Capsules taken orally once per day for 28 days
  Interventions: Drug: TZP-102

INTERVENTIONS:
Drug: TZP-102
  Arms: 10 mg TZP-102; 20 mg TZP-102; 40 mg TZP-102
Drug: Placebo
  Arms: 10 mg TZP-102; 20 mg TZP-102; Placebo

SUMMARY:
The purpose of this study is to evaluate the effect of TZP-102 on gastric emptying rate, gastroparesis symptoms and health-related quality of life in diabetic patients with gastroparesis.

ELIGIBILITY:
Inclusion Criteria:

* 18 to 80 years of age, inclusive.
* Type 1 or type 2 diabetes mellitus.
* Female patients of childbearing potential must have a negative serum pregnancy test and use (and agree to continue to use throughout the study) an acceptable method of contraception.
* HbA1c level less than/equal to 10.0 % at the Screening Visit.
* Diagnosis of gastroparesis including (all three of the following requirements apply): i. Documented delayed gastric emptying; ii. A greater than 3 month history of symptoms of gastroparesis; iii. A GCSI Total Score greater than/equal to 2.66 at the Screening Visit and greater than/equal to 1.90 at the Day 1 visit.
* Upper gastrointestinal obstruction ruled out by endoscopy or barium scan.
* Concomitant medications must be stable for at least 2 weeks leading up to the Baseline Visit and be maintained during the study.
* Body Mass Index (BMI) < 35.
* Delayed gastric emptying by breath test demonstrated at the Baseline Visit.

Exclusion Criteria:

* Persistent daily vomiting
* Gastrectomy, obesity surgery, fundoplication, or vagotomy/pyloroplasty.
* Pyloric Botox within 6 months prior to Screening Visit.
* NG, PEG or PEJ feeding tube.
* Required in-patient hospitalization for treatment of gastroparesis within 2 weeks prior to the Screening Visit.
* Parenteral nutrition for treatment of gastroparesis within 2 months prior to the Screening Visit.
* Active gastric pacemaker within 3 months prior to the Screening Visit.
* Participation in an investigational study within 30 days prior to study entry.
* Chronic severe diarrhea.
* Diabetic ketoacidosis requiring hospitalization within 30 days prior to study entry.
* History of any eating disorder within 2 years prior to study entry.
* Significant chronic obstructive pulmonary disease or chronic asthma.
* Patient is a heavy smoker, and/or unable or unwilling to abstain from smoking during each of the three study visits during which the gastric emptying breath tests will be performed.
* History of risk factors for Torsades de Pointes.
* Patient requires treatment with certain concomitant medications known to have a clinically recognized risk for Torsades de Pointes.
* History of acute myocardial infarction (MI) or unstable angina within 12 months prior to study entry.
* History of any psychiatric disorder or cognitive impairment that would interfere with participation in the study.
* History of alcohol dependency within 2 years prior to study entry.
* Taking opiates for abdominal pain.
* History of HIV infection.
* History of Hepatitis B or C currently exhibiting symptoms expected to worsen during course of study.
* Requires dialysis or has severely impaired renal function.
* Severe impairment of liver function.
* Uncontrolled hypo- or hyperthyroidism.
* History of adrenal insufficiency.
* Pregnant or is breast-feeding.
* Allergic to or intolerant of wheat, egg, soy or milk products.
* Patient requires a gluten-free diet.
* Any other medical condition or social circumstance that, in the investigator's opinion, makes it inappropriate for the patient to participate in this clinical trial.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 92 (Actual)
Dates: Start 2009-04; Primary Completion 2010-04 (Actual); Study Completion 2010-04 (Actual)

PRIMARY OUTCOMES:
change from baseline in gastric half-emptying time | study days 1 and 28

SECONDARY OUTCOMES:
change from baseline in gastroparesis symptoms and health-related quality of life | study days 8, 15 and 28

CONTACTS AND LOCATIONS:
Locations (23):
- United States (11):
  - Long Beach VA Medical Center, Long Beach, California
  - Impact Clinical Trials, Los Angeles, California
  - California Pacific Medical Center Research Institute, San Francisco, California
  - University of South Florida/Tampa General Hospital, Tampa, Florida
  - Saint John's Research Institute, Anderson, Indiana
  - University of Kansas Medical Center, Kansas City, Kansas
  - Univ. of Louisville Medical-Dental Complex, Louisville, Kentucky
  - Beth Israel Deaconess Medical Center, Boston, Massachusetts
  - Dartmouth Hitchcock Medical Center, Lebanon, New Hampshire
  - Wake Research Associates, Raleigh, North Carolina
  - Texas Tech Univ. Health Sciences Center Dept. of Medicine, El Paso, Texas
- Denmark (4):
  - Aalborg Hospital, Aalborg
  - Aarhus University Hospital, Aarhus
  - Steno Diabetes Center, Gentofte Municipality
  - Odense University Hospital, Odense
- Haukeland University Hospital, Bergen, Norway
- Poland (3):
  - Uniwersytecki Szpital Kliniczny w Bialymstoku, Bialystok
  - Oddzial Kliniczny Diabetologii Samodzielny Publiczny Zaklad, Lodz
  - Samodzielny Publiczny Centralny Szpital Kliniczny w Warszawie, Warsaw
- Karolinska University Hospital, Stockholm, Sweden
- United Kingdom (3):
  - Ipswich Hospital NHS Trust, Ipswich
  - Leicester Royal Infirmary, Leicester
  - Wellcome Truest Clinical Research Facility, Manchester